CLINICAL TRIAL: NCT06273436
Title: Comparing Standard of Care Versus a Technology-Based Approach To Reduce Postpartum Emergency Department Visits
Brief Title: Healing, Equity, Advocacy and Respect for Mamas
Acronym: HEAR4Mamas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Constance Guille, Professor - Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00130902
Record Dates: First submitted 2024-01-27; First posted 2024-02-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Complication
Keywords: AIM (Alliance for Innovation on Maternal Health) safety bundles; Randomized Controlled Trial (RCT); Emergency Department (ED) visits; Shared Decision Making (SDM); Patient-Reported Outcomes (PROs); Patient Stakeholder Group (PSG); Study Advisory Committee (SAC)
MeSH Terms: conditions — Episodic Ataxia, Type 1; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): AIM (AIM Alliance for Innovation on Maternal Health) safety bundles delivered in-person
- Usual Care plus H.E.A.R. for Mamas (Experimental): H.E.A.R. for Mamas is designed to provide the AIM (Alliance for Innovation on Maternal Health) Postpartum Discharge Transition education systematically and to frequently monitor women for signs and symptoms of postpartum complications using simple, patient-centered technology (text/phone).
  Interventions: Other: H.E.A.R. for Mamas

INTERVENTIONS:
Other: H.E.A.R. for Mamas — H.E.A.R. for Mamas is a patient and provider informed, multicomponent intervention that uses simple text/phone-based screenings to systematically and frequently monitor women for postpartum complications, chronic conditions and SDoH (Social Determinants of Health) and provides patients with immediate feedback and recommendations based on their screenings.
  Arms: Usual Care plus H.E.A.R. for Mamas

SUMMARY:
The goal of the proposed research is to test the comparative effectiveness of AIM safety bundles for post-partum women delivered in-person vs. via text/phone to improve early detection of and timely care for complications during the first six weeks postpartum for women experiencing significant health disparities.

DETAILED DESCRIPTION:
The purpose of the study is to learn if a program for newborn mom's can improve detection of complications after delivery and help women get medical care quickly and easily. Participants will be asked to complete a survey at the time of enrollment and at 3 additional times. All surveys can be completed via cell-phone or email. All women will be followed for 1-year after delivery. Women that enroll will be assigned to one of two groups: usual in person care OR usual in-person care PLUS a text message-based program that will ask about sign and symptoms of complications that may occur after delivery. If there is a concern, a nurse advocate will call on the phone to discuss options and help refer to care if needed. Participants will be paid for their time in completing surveys.

ELIGIBILITY:
Inclusion Criteria for Postpartum Women

* Postpartum woman within approximately 2 weeks of delivering a baby of gestational age ≥ 26 weeks in South Carolina.
* Aged 16-49 years old.
* Insured by Medicaid.

Exclusion Criteria for Postpartum Women

* Plans to relocate outside of SC anytime during the postpartum year.
* Plans to discontinue Medicaid health insurance during the postpartum year.
* Speaks a language other than English or Spanish.
* Incarcerated/pending incarceration during peripartum period.
* Currently institutionalized.
* Enrolled in current MUSC study funded by PCORI (#Pro00123833)
* Does not have and/or does not wish to use their personal cell phone for the study.

Inclusion Criteria for Obstetric Providers and Hospital Administrators

- OB provider working at a delivery hospital in SC and directly involved in the care of postpartum women; or hospital administrator working in a delivery hospital in SC and job responsibilities relate to the postpartum unit.

Exclusion Criteria for Obstetric Providers and Hospital Administrators

* Less than 1 month of HEAR 4 Mamas experience if involved in the hospital where participants are recruited from.
* Unable or unwilling to commit to completing surveys or an interview.
* Speaking a language other than English.

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Postpartum woman within approximately 2 weeks of delivery Aged 16-49 years old.
Enrollment: 2894 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Emergency Department (ED) visits within six weeks postpartum | Within six weeks following the delivery
  Percent of postpartum women with an ED visit that occurs within six weeks following delivery

SECONDARY OUTCOMES:
Patient Reported Outcomes (PROs) | time of study enrollment (baseline=0), and 3, 6, and 12 months postpartum
  Secondary outcomes will include PROs which will be measured at the time of study enrollment (baseline=0), and 3, 6, and 12 months postpartum.

OTHER OUTCOMES:
Social Determinants of Health (SDoH), Patient Activation, Shared Decision Making | HRSN, PAM-10, and SDM-Q-9 will be measured at study enrollment (baseline=0), 3, 6, and 12 months postpartum
  SDoH will be measured by the Accountable Health Communities-Health-Related Social Needs (HRSN) and includes assessment of economic instability, low social support, food scarcity etc.
Patient Activation | HRSN, PAM-10, and SDM-Q-9 will be measured at study enrollment (baseline=0), 3, 6, and 12 months postpartum
  Patient activation will be measured by the Patient Activation Measure (PAM-10).
Shared Decision Making | HRSN, PAM-10, and SDM-Q-9 will be measured at study enrollment (baseline=0), 3, 6, and 12 months postpartum
  Perception of the shared decision-making process will be measured by Shared Decision-Making Questionnaire (SDM-Q-9).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States